CLINICAL TRIAL: NCT01007929
Title: An Open-Label. Phase I Study to Assess the Excretion of Radioactivity, Metabolic Profiles and Pharmacokinetics Following a Single Oral Dose of 60 mg of [14C] AZD1236 in Healthy Male Subjects
Brief Title: Open-Label Absorption, Distribution, Metabolism, Excretion (ADME) and Pharmacokinetics (PK) Following a Single Oral Dose of AZD1236 in Healthy Male Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Future development of AZD1236 is currently under review by the project team and no new studies will be started until this review is completed.
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4260C00010
Record Dates: First submitted 2009-10-29; First posted 2009-11-05 (Estimated); Last update posted 2009-11-20 (Estimated); Status verified 2009-11

CONDITIONS: Healthy
Keywords: ADME; safety; oral solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): 14C-AZD1236
  Interventions: Drug: 14C-AZD1236

INTERVENTIONS:
Drug: 14C-AZD1236 — Oral solution 1mg/mL

SUMMARY:
The purpose of this study is to characterise the metabolism, excretion and pharmacokinetics of a single oral dose of [14C] AZD1236 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Non-smokers

Exclusion Criteria:

* Subjects who are exposed to radiation exposure as part of their occupation
* Subjects exposed to radiation levels above background of >5 mSv in last year, >10 mSv over last 5 years or a cumulative total of > 1 mSv per year of life
* A history or presence of conditions known to interfere with the absorption, distribution, metabolism or excretion for drugs eg. haematological, gastrointestinal, hepatic or renal disease etc

Ages: 50 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2009-10; Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic profile. Concentration of AZD1236 in plasma | Before and after dosing
Total Radioactivity | Before and after dosing

SECONDARY OUTCOMES:
Adverse events, clinical chemistry, haematology, urinalysis, pulse and blood pressure, ECG and physical examination | Before and after dosing

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca CPU Medical Director, Principal Investigator — AstraZeneca
Locations (1):
- Research Site, Macclesfield, CHESHIRE, United Kingdom